CLINICAL TRIAL: NCT04907890
Title: Long Term Outcomes in COVID-19 Patients Recruited in the CORIST Project: Longitudinal Data and Case-control Study
Brief Title: Long Term Outcomes in COVID-19 Patients Recruited in the CORIST Project
Acronym: CORIST-2
Status: Withdrawn | Type: Observational
Why Stopped: Severe difficulties in enrolling individuals
Sponsor: Neuromed IRCCS (Other)
Collaborators: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Augusto Di Castelnuovo, Principal Investigator, Neuromed IRCCS
Other Study IDs: DEP_012021
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Sars-CoV-2 Infection; Long Covid19
Keywords: Sars-CoV-2; Long Covid19; Case-control study
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: All survivor patients hospitalised for COVID-19 and previously recruited in the CORIST study
- Controls 1: Individuals who had a positive diagnosis for SARS-Cov-2 infection in the past (at least 6 months) and that was never hospitalised for COVID-19 as he/she had not severe symptoms.
- Controls 2: Individuals who was never diagnosed for SARS-Cov-2 infection

SUMMARY:
Months after seemingly recovering from COVID-19, many patients continue to suffer from major long-term effects. Interestingly, the existence of direct link between the severity of the disease in its acute phase and the severity of the long-lasting symptoms is uncertain. We aim at characterizing the long term outcomes in patients hospitalised for COVID-19 including symptoms, medical history, persistent organ damage and neurological and behavioural sequelae.

DETAILED DESCRIPTION:
The aims of this project are: 1) to estimate the degree of physical disability, including psychological sequelae, in survivors of COVID-19 >1-year post hospital discharge and how these long term effect are related to COVID-19 or Sars-Cov-2 infection; 2) to assess if a link between the severity or the treatment of the disease in its acute phase and the severity of the long-lasting symptoms exists.

Aims will be accomplished by using data from the COVID-19 RISK and Treatments (CORIST) Project (ClinicalTrials.gov ID: NCT04318418). The CORIST study included N=4,396 patients hospitalized for SARS-Cov-2 infection in 35 hospitals across Italy, between February 2020 and May 2020. Within each participating hospital, clinical data were abstracted from electronic medical records. Collected data included patients' demographics, laboratory tests, medications in use, history of disease and prescribed pharmacological therapy for COVID-19 treatment. Information on the most severe manifestation of COVID-19 occurred during hospitalization was also captured.

All survivor patients previously recruited in the CORIST study (N=3,648), will be reached by phone by the hospital in which they were healed for COVID-19, informed about the research objectives and procedure and, if they will accept to participate, they will ask to sign an institutional review board consent electronic form. Participants will be requested to return a series of web-based, validated questionnaires aimed at evaluating: 1) occurrence of COVID-19-related symptoms such as fatigue, dizziness, etc.; 2) behavioural features and modifications (e.g., disturbances in sleep, vision, hearing or olfaction); 3) neuropsychological evaluation, regarding multiple cognitive domains (e.g. memory domain, motivational factors, emotional state assessment, mood disturbance and quality of life); 4) change in dietary habits.

Aim 1 Each participant ("case") will be asked to select two control subjects with the following characteristics: control1) same sex, ±5 years, who had a positive diagnosis for SARS-Cov-2 infection in the past (at least 6±2 months) and that was never hospitalised for COVID-19 as he/she had not severe symptoms and control2) same sex, ±5 years, who was never diagnosed for SARS-Cov-2 infection. Each accepting control will be asked to return similar (appropriately modified) questionnaires as cases. Comparisons of cases with control1 individuals will offer evidence of long-term effects due to severity of COVID-19, whereas contrasts of cases or control1 with control2 persons will give indication of long-term effects due to SARS-Cov-2 infection, irrespective from COVID-19.

Aim 2 We expect that a large proportion of case patients has undergone a medical visit in the months after recovering by COVID-19, in the same hospital in which they were healed. For these patients, all available medical information (data on fibrosis, dyspnoea, thoracic pain, respiratory, cardiac, neurological and psychiatric diseases) gathered at follow-up visit will be collected. This bulk of information, together with that attained from questionnaires as described in aim 1 will be related to data (already available to us) from CORIST project and will allow test if a link between the severity or the management in hospital of the disease in its acute phase and the severity of the long-lasting symptoms exists.

ELIGIBILITY:
Inclusion Criteria:

cases: survivor patients previously recruited in the CORIST study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: survivor patients previously recruited in the CORIST study Each case will be asked to select two control subjects with the following characteristics: control1) same sex, ±5 years, who had a positive diagnosis for SARS-Cov-2 infection in the past (at least 6 months) and that was never hospitalised for COVID-19 as he/she had not severe symptoms and control2) same sex, ±5 years, who was never diagnosed for SARS-Cov-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Medical symptoms | 1 year
  Occurrence of COVID-19-related medical symptoms

SECONDARY OUTCOMES:
Difference between cases and controls in behavioural features as assessed by PHQ-9 Depression Test Questionnaire | 1 year
  Differences will be evaluated contrasting cases with both two types of controls and comparing the two groups of controls each other
Difference between cases and controls in physicological features as assessed by GAD7 Anxiety Test Questionnaire | 1 year
  Differences will be evaluated contrasting cases with both two types of controls and comparing the two groups of controls each other
Difference between cases and controls in physicological features as assessed by the Psychological resilience Test (CONNOR-DAVIDSON - 10 items) | 1 year
  Differences will be evaluated contrasting cases with both two types of controls and comparing the two groups of controls each other
Difference between cases and controls in dietary habits as assessed by the mediterranean diet adherence score | 1 year
  Differences will be evaluated contrasting cases with both two types of controls and comparing the two groups of controls each other

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Department of Epidemiology and Prevention, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] COVID-19 RISK and Treatments (CORIST) Collaboration. Use of hydroxychloroquine in hospitalised COVID-19 patients is associated with reduced mortality: Findings from the observational multicentre Italian CORIST study. Eur J Intern Med. 2020 Dec;82:38-47. doi: 10.1016/j.ejim.2020.08.019. Epub 2020 Aug 25. PMID 32859477
- [Result] Di Castelnuovo A, Bonaccio M, Costanzo S, Gialluisi A, Antinori A, Berselli N, Blandi L, Bruno R, Cauda R, Guaraldi G, My I, Menicanti L, Parruti G, Patti G, Perlini S, Santilli F, Signorelli C, Stefanini GG, Vergori A, Abdeddaim A, Ageno W, Agodi A, Agostoni P, Aiello L, Al Moghazi S, Aucella F, Barbieri G, Bartoloni A, Bologna C, Bonfanti P, Brancati S, Cacciatore F, Caiano L, Cannata F, Carrozzi L, Cascio A, Cingolani A, Cipollone F, Colomba C, Crisetti A, Crosta F, Danzi GB, D'Ardes D, de Gaetano Donati K, Di Gennaro F, Di Palma G, Di Tano G, Fantoni M, Filippini T, Fioretto P, Fusco FM, Gentile I, Grisafi L, Guarnieri G, Landi F, Larizza G, Leone A, Maccagni G, Maccarella S, Mapelli M, Maragna R, Marcucci R, Maresca G, Marotta C, Marra L, Mastroianni F, Mengozzi A, Menichetti F, Milic J, Murri R, Montineri A, Mussinelli R, Mussini C, Musso M, Odone A, Olivieri M, Pasi E, Petri F, Pinchera B, Pivato CA, Pizzi R, Poletti V, Raffaelli F, Ravaglia C, Righetti G, Rognoni A, Rossato M, Rossi M, Sabena A, Salinaro F, Sangiovanni V, Sanrocco C, Scarafino A, Scorzolini L, Sgariglia R, Simeone PG, Spinoni E, Torti C, Trecarichi EM, Vezzani F, Veronesi G, Vettor R, Vianello A, Vinceti M, De Caterina R, Iacoviello L; COvid-19 RISk and Treatments (CORIST) collaboration. Common cardiovascular risk factors and in-hospital mortality in 3,894 patients with COVID-19: survival analysis and machine learning-based findings from the multicentre Italian CORIST Study. Nutr Metab Cardiovasc Dis. 2020 Oct 30;30(11):1899-1913. doi: 10.1016/j.numecd.2020.07.031. Epub 2020 Jul 31. PMID 32912793
- [Result] Di Castelnuovo A, Costanzo S, Antinori A, Berselli N, Blandi L, Bonaccio M, Cauda R, Guaraldi G, Menicanti L, Mennuni M, Parruti G, Patti G, Santilli F, Signorelli C, Vergori A, Abete P, Ageno W, Agodi A, Agostoni P, Aiello L, Al Moghazi S, Arboretti R, Astuto M, Aucella F, Barbieri G, Bartoloni A, Bonfanti P, Cacciatore F, Caiano L, Carrozzi L, Cascio A, Ciccullo A, Cingolani A, Cipollone F, Colomba C, Colombo C, Crosta F, Danzi GB, D'Ardes D, de Gaetano Donati K, Di Gennaro F, Di Tano G, D'Offizi G, Fantoni M, Fusco FM, Gentile I, Gianfagna F, Grandone E, Graziani E, Grisafi L, Guarnieri G, Larizza G, Leone A, Maccagni G, Madaro F, Maitan S, Mancarella S, Mapelli M, Maragna R, Marcucci R, Maresca G, Marongiu S, Marotta C, Marra L, Mastroianni F, Mazzitelli M, Mengozzi A, Menichetti F, Meschiari M, Milic J, Minutolo F, Molena B, Montineri A, Mussini C, Musso M, Niola D, Odone A, Olivieri M, Palimodde A, Parisi R, Pasi E, Pesavento R, Petri F, Pinchera B, Poletti V, Ravaglia C, Rognoni A, Rossato M, Rossi M, Sangiovanni V, Sanrocco C, Scorzolini L, Sgariglia R, Simeone PG, Taddei E, Torti C, Vettor R, Vianello A, Vinceti M, Virano A, Vocciante L, De Caterina R, Iacoviello L. Heparin in COVID-19 Patients Is Associated with Reduced In-Hospital Mortality: The Multicenter Italian CORIST Study. Thromb Haemost. 2021 Aug;121(8):1054-1065. doi: 10.1055/a-1347-6070. Epub 2021 Feb 28. PMID 33412596
- [Result] COVID-19 RISk and Treatments (CORIST) Collaboration. RAAS inhibitors are not associated with mortality in COVID-19 patients: Findings from an observational multicenter study in Italy and a meta-analysis of 19 studies. Vascul Pharmacol. 2020 Dec;135:106805. doi: 10.1016/j.vph.2020.106805. Epub 2020 Sep 28. PMID 32992048
- [Result] Di Castelnuovo A, De Caterina R, de Gaetano G, Iacoviello L. Controversial Relationship Between Renin-Angiotensin System Inhibitors and Severity of COVID-19: Announcing a Large Multicentre Case-Control Study in Italy. Hypertension. 2020 Aug;76(2):312-313. doi: 10.1161/HYPERTENSIONAHA.120.15370. Epub 2020 May 8. No abstract available. PMID 32383624
- [Result] Ruggiero E, Mignogna C, Costanzo S, Persichillo M, Di Castelnuovo A, Esposito S, Cerletti C, Donati MB, de Gaetano G, Iacoviello L, Bonaccio M; Moli-LOCK Study Investigators. Changes in the consumption of foods characterising the Mediterranean dietary pattern and major correlates during the COVID-19 confinement in Italy: results from two cohort studies. Int J Food Sci Nutr. 2021 Dec;72(8):1105-1117. doi: 10.1080/09637486.2021.1895726. Epub 2021 Apr 6. PMID 33823720
- [Result] Bonaccio M, Costanzo S, Ruggiero E, Persichillo M, Esposito S, Olivieri M, Di Castelnuovo A, Cerletti C, Donati MB, de Gaetano G, Iacoviello L; Moli-LOCK Study Investigators. Changes in ultra-processed food consumption during the first Italian lockdown following the COVID-19 pandemic and major correlates: results from two population-based cohorts. Public Health Nutr. 2021 Aug;24(12):3905-3915. doi: 10.1017/S1368980021000999. Epub 2021 Mar 5. PMID 33663640